CLINICAL TRIAL: NCT02831348
Title: Association of Transcutaneous Pulse CO-oximetry With Inflammatory Lung Diseases
Acronym: COOX
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan M. Gaffin, Principal Investigator, Boston Children's Hospital
Other Study IDs: ChildrenH
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Asthma; Allergic Rhinitis; Cystic Fibrosis; Pneumonia
Keywords: Asthma; Allergic rhinitis; Rhinitis; Pneumonia; Cystic fibrosis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Cystic Fibrosis; Pneumonia; Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Uncontrolled asthma: Indicated by an asthma control test (ACT) score of <20 and asthma symptoms of cough, wheeze, or chest tightness for more than 2 days in the prior 2 weeks, OR current asthma exacerbation indicated by the prescription of a short course (3-5 days) of systemic corticosteroids by treating provider at the time of visit.
- Controlled asthma: Indicated by an ACT score of >19, or spirometry results within 10% of year's best value (based on FEV1).
- Pneumonia: Indicated by an admission diagnosis of pneumonia with chest X-ray consistent with the diagnosis, based on attending radiologist's interpretation.
- Controlled allergic rhinitis: Indicated by a rhinitis control assessment test (RCAT) score of >= 21.
- Uncontrolled allergic rhinitis: Indicated by an RCAT score of <21.
- Cystic fibrosis (exacerbated): Indicated by treating physician's assessment of cystic fibrosis respiratory exacerbation within 24 hours of initial antibiotic therapy.
- Cystic fibrosis (stable): Indicated by diagnosis of cystic fibrosis with baseline symptoms and with spirometry results (based on FEV1) within 5% of year's best value.
- Control: Indicated by a negative history of any of the conditions characterizing the other groups.

SUMMARY:
This is a pilot cross-sectional study of measured transcutaneous CO-oximetry in children with inflammatory and non-inflammatory conditions.

DETAILED DESCRIPTION:
Children and young adults age 6-24 with the following conditions: asthma, pneumonia, allergic rhinitis, cystic fibrosis, and well child (without inflammatory illness) will be recruited.

Subjects will be asked to complete a brief screening survey to determine if they meet inclusion criteria. Enrolled subjects will be asked to complete questionnaire forms to characterize their health, current symptoms, medications, and common exposures. Transcutaneous carboxyhemoglobin will be recorded.

This study is cross-sectional and will only require one visit coinciding with the clinical visit. Analysis will determine the pairwise differences in SpCO between conditions tested.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of asthma, pneumonia, allergic rhinitis, or none of the previous (control group)
* Ability to complete study procedures

Exclusion Criteria:

* Cardiopulmonary disease outside of the specific conditions for inclusion
* Prematurity
* Congenital heart disease
* Current diagnosis of more than one of the following: asthma, pneumonia, allergic rhinitis, cystic fibrosis, or - for controls - any current infection
* Recent serious bacterial infection (except for pneumonia in the pneumonia group)
* Concurrent clinical chest X-ray with findings other those that expected for the group (i.e. normal chest X-ray in pneumonia group or suspected pneumonia on chest X-ray in asthma group). To be determined by attending radiologist's interpretation.

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Age range 6-24years old. All genders, races, and ethnicities were sampled, provided they could complete the study requirements.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
SpCO comparison: uncontrolled asthma v. other groups | Time of visit
  A pairwise comparison of mean SpCO will be performed between asthma exacerbation group and each other group, e.g., asthma exacerbation v. stable asthma, asthma exacerbation v. pneumonia, etc. An independent t-test will be used to determine statistical significance of the difference of means.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gaffin, MD. MMSc., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No